CLINICAL TRIAL: NCT01048775
Title: Investigation on the Diagnostic and Predictive Value of Bilateral Bispectral Index (BIS)-Monitoring in Cardiac Surgery
Brief Title: Bilateral Bispectral Index (BIS)-Monitoring in Cardiac Surgery Patients
Status: Completed | Type: Observational
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Martin Soehle, Consultant of Anaesthesiology, University Hospital, Bonn
Other Study IDs: BLB-09; Projekt-Nr UKB: N-017.0160
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Last update posted 2012-04-17 (Estimated); Status verified 2012-04

CONDITIONS: Cardiac Surgery Patients
Keywords: bispectral index; cardiac surgery; asymmetry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The bispectral index (BIS) is derived from a single-channel electroencephalogram (EEG) and provides information on the anaesthetic depth. Recently, a bilateral two-channel EEG-sensor has been introduced to monitor the BIS on both cerebral hemispheres. In some patients significant left-right differences may occur, whereas no relevant side differences are expected in the majority of patients.

The aim of this study is to

* investigate the incidence, duration and degree of left-right BIS differences
* examine the relation between BIS differences and occurrence of cognitive deficits

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for cardiac surgery

Exclusion Criteria:

* pregnancy

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients treated at a University Hospital
Sampling Method: Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2010-02

PRIMARY OUTCOMES:
BIS side difference | intra- and postoperative (day 1)

SECONDARY OUTCOMES:
ADL = Activity of Daily Living | 6 month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Martin Soehle, M.D., D.E.S.A., D. habil., Principal Investigator — Dept of Anaesthesiology and Intensive Care Medicine
Locations (1):
- Dept. of Anaesthesiology and Intensive Care Medicine, University of Bonn, Bonn, Germany

REFERENCES:
- [Derived] Soehle M, Dittmann A, Ellerkmann RK, Baumgarten G, Putensen C, Guenther U. Intraoperative burst suppression is associated with postoperative delirium following cardiac surgery: a prospective, observational study. BMC Anesthesiol. 2015 Apr 28;15:61. doi: 10.1186/s12871-015-0051-7. PMID 25928189